CLINICAL TRIAL: NCT01437397
Title: A Phase III, Randomized, Double-blind, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Tolerability of Two Fixed Dose Combinations of Aclidinium Bromide/Formoterol Fumarate Compared With Aclidinium Bromide, Formoterol Fumarate and Placebo for 24- Weeks Treatment in Patients With Moderate to Severe, Stable Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Efficacy, Safety and Tolerability of Aclidinium Bromide/Formoterol Fumarate Compared With Aclidinium Bromide and Formoterol Fumarate in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAC-MD-31
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Aclidinium/formoterol Fixed Dose Combination (FDC) 400/12μg
  Interventions: Drug: Aclidinium Bromide/Formoterol Fumarate
- 2 (Experimental): Aclidinium/formoterol Fixed Dose Combination (FDC) 400/6μg
  Interventions: Drug: Aclidinium Bromide/Formoterol Fumarate
- 3 (Active Comparator): Aclidinium monotherapy 400 μg
  Interventions: Drug: Aclidinium Bromide
- 4 (Active Comparator): Formoterol monotherapy 12 μg
  Interventions: Drug: Formoterol Fumarate
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium Bromide/Formoterol Fumarate — Inhaled Aclidinium/formoterol FDC 400/12μg, twice per day
  Arms: 1
Drug: Aclidinium Bromide/Formoterol Fumarate — Inhaled Aclidinium/formoterol FDC 400/6μg, twice per day
  Arms: 2
Drug: Aclidinium Bromide — Inhaled Aclidinium 400 μg, twice per day
  Arms: 3
Drug: Formoterol Fumarate — Inhaled Formoterol 12 μg, twice per day
  Arms: 4
Drug: Placebo — Inhaled dose-matched placebo, twice per day
  Arms: 5

SUMMARY:
The purpose of this Phase III study is to assess the maintenance bronchodilator effects of the fixed dose combination versus monotherapies. This study will also assess the effects of the fixed dose combination in terms of COPD symptoms, disease related health status and the long-term safety and tolerability of the fixed dose combination. This study will include a 24 week treatment period, preceding by a run-in period, followed by a two week follow up visit. All patients will be randomized to one of four treatment arms or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 40 years of age
* Current or former cigarette smoker with a cigarette smoking history of at least 10 pack-years
* A diagnosis of stable moderate to severe COPD and stable airway obstruction as defined by the GOLD guidelines and stable airway obstruction. Patients had to have a postbronchodilator FEV1/FVC ratio < 70% at Visit 1 (GOLD, 2010)
* Post-albuterol/salbutamol FEV1 values ≥ 30% and < 80% of predicted value. FEV1 was measured at the Screening Visit (Visit 1) 10 to 15 minutes after inhalation of albuterol/salbutamol. Predicted normal used for calculation purposes were based on National Health and Nutrition Examination Survey III predicted values (Hankinson et al, 1999)
* Able to perform acceptable and repeatable pulmonary function testing for FEV1 according to ATS/ERS criteria (Miller et al, 2005) at Screening Visit (Visit 1) and throughout their participation in the trial
* Negative serum β-human chorionic gonadotropin pregnancy test at Visit 1 and must have been using hormonal contraceptives or a barrier method plus a spermicidal agent; otherwise at least 1-year postmenopausal or surgically sterile, defined as having a hysterectomy or tubal ligation (applied to female patients only)
* Judged by the Principal Investigator to be in otherwise good stable health based on medical history, physical examination, ECGs, and routine laboratory data evaluations
* Patients previously randomized in an aclidinium monotherapy trial were permitted as long as it had been at least 6 months since the completion of their previous trial participation
* Able to understand the study procedures and be willing to participate in the study as indicated by signing the informed consent

Exclusion Criteria:

* Hospitalization for an acute COPD exacerbation within 3 months before Visit 1
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the 6 weeks before Visit 1. Patients who developed a respiratory tract infection or COPD exacerbation during the washout or run-in period were discontinued from the study before randomization
* Any clinically significant respiratory conditions other than COPD, including active tuberculosis, history of interstitial lung disease, pulmonary thromboembolic disease, history of α1-antitrypsin deficiency, pulmonary resection, lung volume surgery, or any other thoracic surgery during the past 12 months, history of bronchiectasis secondary to respiratory diseases other than COPD (eg, cystic fibrosis, Kartagener syndrome), post organ transplantation, or expected to require thoracotomy or other lung surgery during the study
* Clinical history suggesting that the patient had asthma as opposed to COPD (Study Physician was to be contacted to discuss eligibility, if necessary)
* Chronic use of oxygen therapy ≥ 15 hours/day
* Body mass index(BMI) ≥ 40 kg/m2
* Patients who intended to start a pulmonary rehabilitation program during the trial were excluded, as well as those who finished or started it within 3 months prior to Screening Visit
* Clinically significant cardiovascular conditions including: myocardial infarction within the previous 6 months; newly diagnosed arrhythmia within the previous 3 months; unstable angina; unstable arrhythmia that had required changes in pharmacological therapy or other intervention within the previous 6 months; the presence of an automated implantable cardioverter-defibrillator; history of thoracic surgery within the past year before screening; hospitalization within the previous 12 months for heart failure of New York Heart Association functional class III (marked limitation of physical activity and only comfortable at rest, less than ordinary activity causes fatigue, palpitation or dyspnea), or class IV (unable to carry out any physical activity without discomfort) (Criteria Committee of the New York Heart Association criteria, 1994)
* Any uncontrolled infection that may have placed the patient at risk resulting from human immunodeficiency virus, active hepatitis and/or patients with diagnosed active tuberculosis
* QTcB > 470 msec in the resting ECGs performed at Screening (Visit 1), as indicated in the centralized ECG vendor generated report. Patients who were on a stable dose of medication that may prolong the QTc, but had a documented, stable, and normal QTc, could have been considered
* QTcB > 470 msec in the resting ECGs performed before randomization at Visit 2, as indicated in the paper tracing generated by the Sponsor-provided ECG equipment
* Clinically relevant abnormalities in the results of the clinical laboratory tests, in ECG parameters other than QTc, or in the physical examination or vital signs at Visit 1 except for those related to COPD
* History of drug or alcohol abuse within the previous 5 years
* Any other serious or uncontrolled physical or mental condition/disease that, as judged by the Investigator, could have placed the patient at higher risk derived from his/her participation in the study, could have confounded the results of the study, or would be likely to have prevented the patient from complying with the requirements of the study or completing the study. If there was a history of such disease, but the condition had been stable for more than 1 year and was judged by the Investigator not to interfere with the patient's participation in the study, the patient may have been included, with the documented approval of the Study Physician
* History of hypersensitivity reaction to inhaled anticholinergics, beta-2 agonists, sympathomimetic amines, or inhaled medication or any component thereof (including report of paradoxical bronchospasm) or a history of acute urinary retention, symptomatic benign prostatic hyperplasia, bladder neck obstruction, or narrow-angle glaucoma. (Note: Patients who had well controlled, stable, asymptomatic benign prostatic hyperplasia were not to be excluded)
* Sitting, resting systolic BP ≥ 160 mm Hg and/or diastolic BP ≥ 100 mm Hg at Visit 1 and Visit 2
* Unable to use a multidose dry-powder inhaler or a pressurized metered-dose inhaler
* Treatment with any other investigational product within 30 days (or 6 half-lives, whichever was longer) before Visit 1
* Previous participation in a clinical trial with aclidinium bromide in an FDC therapy
* Pregnant or breastfeeding
* Current diagnosis of cancer (present in the patient) other than basal or squamous cell skin cancer. Patients who had a history of cancer must have been cleared before Visit 1 (Screening) on a case-by-case basis
* Patients who did not maintain regular day/night, waking/sleeping cycles (eg, night shift workers)
* Patients who intended to use any concomitant medication not permitted by this protocol or who had not undergone the required washout period for a particular prohibited medication (Appendix III of the protocol, which can be found in Appendix 16.1.1 of this report)
* Patients who were unlikely to be compliant with study requirements (eg, take their medication, complete their electronic diaries, attend clinic at the required times)
* Patients who were employees or relatives of employees of the investigative study center, FRI, Almirall, SA, or Pharmaceutical Product Development (PPD, Inc.)
* Patients who had any other conditions that, in the Investigator's opinion, might have indicated the patient to be unsuitable for the study or supported excluding the patient from the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1692 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (222):
- United States (193):
  - Forest Investigative Site 1827, Anniston, Alabama
  - Forest Investigative Site 1920, Athens, Alabama
  - Forest Investigative Site 1162, Birmingham, Alabama
  - Forest Investigative Site 1493, Birmingham, Alabama
  - Forest Investigative Site 1937, Birmingham, Alabama
  - Forest Investigative Site 1893, Florence, Alabama
  - Forest Investigative Site 1824, Gulf Shores, Alabama
  - Forest Investigative Site 2088, Jasper, Alabama
  - Forest Investigative Site 1918, Scottsboro, Alabama
  - Forest Investigative Site 0909, Glendale, Arizona
  - Forest Investigative Site 1958, Mesa, Arizona
  - Forest Investigative Site 1379, Phoenix, Arizona
  - Forest Investigative Site 1822, Anaheim, California
  - Forest Investigative Site 1483, Buena Park, California
  - Forest Investigative Site 1809, Fountain Valley, California
  - Forest Investigative Site 1156, Fresno, California
  - Forest Investigative Site 1871, Lincoln, California
  - Forest Investigative Site 1873, Los Angeles, California
  - Forest Investigative Site 2064, Riverside, California
  - Forest Investigative Site 1427, Sacramento, California
  - Forest Investigative Site 1866, Sacramento, California
  - Forest Investigative Site 1125, San Diego, California
  - Forest Investigative Site 1898, San Diego, California
  - Forest Investigative Site 2009, San Diego, California
  - Forest Investigative Site 1374, Torrance, California
  - Forest Investigative Site 1813, Tustin, California
  - Forest Investigative Site 1883, Vista, California
  - Forest Investigative Site 1380, Golden, Colorado
  - Forest Investigative Site 1137, Pueblo, Colorado
  - Forest Investigative Site 1327, Wheat Ridge, Colorado
  - Forest Investigative Site 1976, Waterbury, Connecticut
  - Forest Investigative Site 1821, Bay Pines, Florida
  - Forest Investigative Site 1154, Brandon, Florida
  - Forest Investigative Site 1944, Brandon, Florida
  - Forest Investigative Site 1364, Clearwater, Florida
  - Forest Investigative Site 1152, Clearwater, Florida
  - Forest Investigative Site 1875, Clearwater, Florida
  - Forest Investigative Site 0670, DeLand, Florida
  - Forest Investigative Site 1516, Edgewater, Florida
  - Forest Investigative Site 0990, Fort Lauderdale, Florida
  - Forest Investigative Site 1513, Hialeah, Florida
  - Forest Investigative Site 1854, Hialeah, Florida
  - Forest Investigative Site 1882, Hollywood, Florida
  - Forest Investigative Site 1543, Jacksonville, Florida
  - Forest Investigative Site 1416, Kissimmee, Florida
  - Forest Investigative Site 1167, Melbourne, Florida
  - Forest Investigative Site 1868, Miami, Florida
  - Forest Investigative Site 1432, Miami, Florida
  - Forest Investigative Site 1979, Miami, Florida
  - Forest Investigative Site 1819, Naples, Florida
  - Forest Investigative Site 1808, North Miami Beach, Florida
  - Forest Investigative Site 1950, Oldsmar, Florida
  - Forest Investigative Site 1145, Ormond Beach, Florida
  - Forest Investigative Site 1094, Panama City, Florida
  - Forest Investigative Site 1803, Pembroke Pines, Florida
  - Forest Investigative Site 974, Pensacola, Florida
  - Forest Investigative Site 1829, Saint Cloud, Florida
  - Forest Investigative Site 1817, Sarasota, Florida
  - Forest Investigative Site 1876, St. Petersburg, Florida
  - Forest Investigative Site 1874, St. Petersburg, Florida
  - Forest Investigative Site 2082, Tamarac, Florida
  - Forest Investigative Site 2053, Tampa, Florida
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1185, Winter Park, Florida
  - Forest Investigative Site 1860, Winter Park, Florida
  - Forest Investigative Site 1982, Albany, Georgia
  - Forest Investigative Site 1900, Atlanta, Georgia
  - Forest Investigative Site 0987, Austell, Georgia
  - Forest Investigative Site 1828, Canton, Georgia
  - Forest Investigative Site 1830, Marietta, Georgia
  - Forest Investigative Site 2089, Woodstock, Georgia
  - Forest Investigative Site 0679, Coeur d'Alene, Idaho
  - Forest Investigative Site 1858, Eagle, Idaho
  - Forest Investigative Site 1095, Normal, Illinois
  - Forest Investigative Site 1912, Normal, Illinois
  - Forest Investigative Site 2051, River Forest, Illinois
  - Forest Investigative Site 2033, Bowling Green, Kentucky
  - Forest Investigative Site 2085, Fort Mitchell, Kentucky
  - Forest Investigative Site 0539, Lexington, Kentucky
  - Forest Investigative Site 1478, Louisville, Kentucky
  - Forest Investigative Site 1519, Owensboro, Kentucky
  - Forest Investigative Site 1811, Covington, Louisiana
  - Forest Investigative Site 1430, New Orleans, Louisiana
  - Forest Investigative Site 1812, Opelousas, Louisiana
  - Forest Investigative Site 1814, Bangor, Maine
  - Forest Investigative Site 1924, Baltimore, Maryland
  - Forest Investigative Site 1865, Hollywood, Maryland
  - Forest Investigative Site 1872, Wheaton, Maryland
  - Forest Investigative Site 1570, Fall River, Massachusetts
  - Forest Investigative Site 1852, Fall River, Massachusetts
  - Forest Investigative Site 1029, North Dartmouth, Massachusetts
  - Forest Investigative Site 1431, North Dartmouth, Massachusetts
  - Forest Investigative Site 1892, Ann Arbor, Michigan
  - Forest Investigative Site 1342, Stevensville, Michigan
  - Forest Investigative Site 1487, Troy, Michigan
  - Forest Investigative Site 1128, Edina, Minnesota
  - Forest Investigative Site 1527, Fridley, Minnesota
  - Forest Investigative Site 2041, Minneapolis, Minnesota
  - Forest Investigative Site 1124, Minneapolis, Minnesota
  - Forest Investigative Site 1619, Plymouth, Minnesota
  - Forest Investigative Site 1118, Rochester, Minnesota
  - Forest Investigative Site 1884, Olive Branch, Mississippi
  - Forest Investigative Site 1587, Chesterfield, Missouri
  - Forest Investigative Site 1602, Kansas City, Missouri
  - Forest Investigative Site 2079, Saint Charles, Missouri
  - Forest Investigative Site 1856, Springfield, Missouri
  - Forest Investigative Site 1867, Springfield, Missouri
  - Forest Investigative Site 1399, St Louis, Missouri
  - Forest Investigative Site 1599, St Louis, Missouri
  - Forest Investigative Site 1831, Bozeman, Montana
  - Forest Investigative Site 1400, Missoula, Montana
  - Forest Investigative Site 1609, Bellevue, Nebraska
  - Forest Investigative Site 1948, Fremont, Nebraska
  - Forest Investigative Site 1815, Lincoln, Nebraska
  - Forest Investigative Site 1363, Omaha, Nebraska
  - Forest Investigative Site 1907, Omaha, Nebraska
  - Forest Investigative Site 1911, Omaha, Nebraska
  - Forest Investigative Site 1908, Omaha, Nebraska
  - Forest Investigative Site 1804, Omaha, Nebraska
  - Forest Investigative Site 1807, Henderson, Nevada
  - Forest Investigative Site 1834, Las Vegas, Nevada
  - Forest Investigative Site 1562, Las Vegas, Nevada
  - Forest Investigative Site 1559, Cherry Hill, New Jersey
  - Forest Investigative Site 1923, Hackensack, New Jersey
  - Forest Investigative Site 1949, Albuquerque, New Mexico
  - Forest Investigative Site 1151, Great Neck, New York
  - Forest Investigative Site 1489, Larchmont, New York
  - Forest Investigative Site 0550, New York, New York
  - Forest Investigative Site 1425, New York, New York
  - Forest Investigative Site 2098, Rochester, New York
  - Forest Investigative Site 1392, Charlotte, North Carolina
  - Forest Investigative Site 2035, Elizabeth City, North Carolina
  - Forest Investigative Site 1366, High Point, North Carolina
  - Forest Investigative Site 1153, Raleigh, North Carolina
  - Forest Investigative Site 1823, Salisbury, North Carolina
  - Forest Investigative Site 1891, Cadiz, Ohio
  - Forest Investigative Site 1134, Canton, Ohio
  - Forest Investigative Site 1885, Cincinnati, Ohio
  - Forest Investigative Site 1806, Cincinnati, Ohio
  - Forest Investigative Site 2028, Cincinnati, Ohio
  - Forest Investigative Site 1903, Cincinnati, Ohio
  - Forest Investigative Site 1361, Columbus, Ohio
  - Forest Investigative Site 1433, Columbus, Ohio
  - Forest Investigative Site 2090, Sylvania, Ohio
  - Forest Investigative Site 1530, Toledo, Ohio
  - Forest Investigative Site 1393, Zanesville, Ohio
  - Forest Investigative Site 1915, Oklahoma City, Oklahoma
  - Forest Investigative Site 1889, Bend, Oregon
  - Forest Investigative Site 2043, Medford, Oregon
  - Forest Investigative Site 1833, Altoona, Pennsylvania
  - Forest Investigative Site 1855, Clairton, Pennsylvania
  - Forest Investigative Site 1820, Downington, Pennsylvania
  - Forest Investigative Site 1423, Erie, Pennsylvania
  - Forest Investigative Site 1899, Langhorne, Pennsylvania
  - Forest Investigative Site 1443, Philadelphia, Pennsylvania
  - Forest Investigative Site 1863, Phoenixville, Pennsylvania
  - Forest Investigative Site 1146, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1449, Tipton, Pennsylvania
  - Forest Investigative Site 1862, Uniontown, Pennsylvania
  - Forest Investigative Site 1832, Cumberland, Rhode Island
  - Forest Investigative Site 1089, East Providence, Rhode Island
  - Forest Investigative Site 2072, Charleston, South Carolina
  - Forest Investigative Site 1905, Charleston, South Carolina
  - Forest Investigative Site 1802, Charleston, South Carolina
  - Forest Investigative Site 1914, Fort Mill, South Carolina
  - Forest Investigative Site 1913, Gaffney, South Carolina
  - Forest Investigative Site 1121, Spartanburg, South Carolina
  - Forest Investigative Site 1957, Brentwood, Tennessee
  - Forest Investigative Site 1526, Fayetteville, Tennessee
  - Forest Investigative Site 1440, Arlington, Texas
  - Forest Investigative Site 1879, Boerne, Texas
  - Forest Investigative Site 1861, Carrollton, Texas
  - Forest Investigative Site 1816, Corsicana, Texas
  - Forest Investigative Site 1890, Dallas, Texas
  - Forest Investigative Site 1332, El Paso, Texas
  - Forest Investigative Site 2012, Fort Worth, Texas
  - Forest Investigative Site 1951, Houston, Texas
  - Forest Investigative Site 1902, Killeen, Texas
  - Forest Investigative Site 1091, McKinney, Texas
  - Forest Investigative Site 1826, Plano, Texas
  - Forest Investigative Site 0526, San Angelo, Texas
  - Forest Investigative Site 1895, San Antonio, Texas
  - Forest Investigative Site 1936, Salt Lake City, Utah
  - Forest Investigative Site 1330, South Burlington, Vermont
  - Forest Investigative Site 1945, Newport News, Virginia
  - Forest Investigative Site 1404, Norfolk, Virginia
  - Forest Investigative Site 1120, Bellingham, Washington
  - Forest Investigative Site 1977, Spokane, Washington
  - Forest Investigative Site 1878, Spokane, Washington
  - Forest Investigative Site 1573, Spokane, Washington
  - Forest Investigative Site 0988, Tacoma, Washington
  - Forest Investigative Site 1870, Tacoma, Washington
  - Forest Investigative Site 1555, Morgantown, West Virginia
- Australia (11):
  - Forest Investigative Site 1991, New Lambton, New South Wales
  - Forest Investigative Site 1987, Redcliffe, Queensland
  - Forest Investigative Site 1973, Woolloongabba, Queensland
  - Forest Investigative Site 1981, Bedford Park, South Australia
  - Forest Investigative Site 1990, Daw Park, South Australia
  - Forest Investigative Site 2251, Toorak Gardens, South Australia
  - Forest Investigative Site 2250, Clayton, Victoria
  - Forest Investigative Site 1972, Fitzroy, Victoria
  - Forest Investigative Site 1986, Geelong, Victoria
  - Forest Investigative Site 1985, Parkville, Victoria
  - Forest Investigative Site 2253, Adelaide, Western Australia
- Canada (10):
  - Forest Investigative Site 1904, Langley, British Columbia
  - Forest Investigative Site 0905, Vancouver, British Columbia
  - Forest Investigative Site 0976, Winnipeg, Manitoba
  - Forest Investigative Site 1877, Sarina, Ontario
  - Forest Investigative Site 1896, Sarnia, Ontario
  - Forest Investigative Site 1171, Toronto, Ontario
  - Forest Investigative Site 2203, Toronto, Ontario
  - Forest Investigative Site 1952, Montreal, Quebec
  - Forest Investigative Site 1859, Québec, Quebec
  - Forest Investigative Site 0943, Saskatoon, Saskatchewan
- New Zealand (8):
  - Forest Investigative Site 1027, Auckland
  - Forest Investigative Site 1970, Christchurch
  - Forest Investigative Site 1967, Dunedin
  - Forest Investigative Site 1964, Dunedin
  - Forest Investigative Site 1968, Hamilton
  - Forest Investigative Site 1965, Tauranga
  - Forest Investigative Site 1980, Tauranga
  - Forest Investigative Site 1025, Wellington

REFERENCES:
- [Derived] Singh D, D'Urzo AD, Donohue JF, Kerwin EM, Molins E, Chuecos F, Ribera A, Jarreta D. An Evaluation Of Single And Dual Long-Acting Bronchodilator Therapy As Effective Interventions In Maintenance Therapy-Naive Patients With COPD. Int J Chron Obstruct Pulmon Dis. 2019 Dec 6;14:2835-2848. doi: 10.2147/COPD.S217710. eCollection 2019. PMID 31827323
- [Derived] Singh D, D'Urzo AD, Chuecos F, Munoz A, Garcia Gil E. Reduction in clinically important deterioration in chronic obstructive pulmonary disease with aclidinium/formoterol. Respir Res. 2017 May 30;18(1):106. doi: 10.1186/s12931-017-0583-0. PMID 28558833
- [Derived] Jones PW, Leidy NK, Hareendran A, Lamarca R, Chuecos F, Garcia Gil E. The effect of aclidinium bromide on daily respiratory symptoms of COPD, measured using the Evaluating Respiratory Symptoms in COPD (E-RS: COPD) diary: pooled analysis of two 6-month Phase III studies. Respir Res. 2016 May 23;17(1):61. doi: 10.1186/s12931-016-0372-1. PMID 27215749
- [Derived] Bateman ED, Chapman KR, Singh D, D'Urzo AD, Molins E, Leselbaum A, Gil EG. Aclidinium bromide and formoterol fumarate as a fixed-dose combination in COPD: pooled analysis of symptoms and exacerbations from two six-month, multicentre, randomised studies (ACLIFORM and AUGMENT). Respir Res. 2015 Aug 2;16(1):92. doi: 10.1186/s12931-015-0250-2. PMID 26233481
- [Derived] D'Urzo AD, Rennard SI, Kerwin EM, Mergel V, Leselbaum AR, Caracta CF; AUGMENT COPD study investigators. Efficacy and safety of fixed-dose combinations of aclidinium bromide/formoterol fumarate: the 24-week, randomized, placebo-controlled AUGMENT COPD study. Respir Res. 2014 Oct 14;15(1):123. doi: 10.1186/s12931-014-0123-0. PMID 25756831
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4060&filename=CSRsynopsis_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 205 sites, 178 in the United States, 9 in Canada, 10 in Australia, and 8 in New Zealand. The first patient was screened in October 2011 and the last patient visit was in February 2013
Pre-assignment Details: A total of 3260 patients were screened for eligibility; 1692 patients were randomized to treatment. A total of 1568 (48.1%) patients screen failed and were discontinued prior to randomization. The primary reason for screening failures was not meeting inclusion/exclusion criteria (41.6%)
Groups:
- Aclidinium/Formoterol 400/12 μg; Aclidinium/Formoterol 400/6 μg: Fixed-dose combination (FDC) administered BID by inhalation
- Aclidinium 400 μg; Formoterol 12 μg; Placebo: Administered BID by inhalation
Period: Overall Study
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Started | 338 | 338 | 340 | 339 | 337
Completed | 272 | 276 | 268 | 270 | 236
Not Completed | 66 | 62 | 72 | 69 | 101
Not completed — Lost to Follow-up | 9 | 4 | 2 | 4 | 5
Not completed — Withdrawal by Subject | 11 | 12 | 24 | 11 | 22
Not completed — Protocol Violation | 10 | 12 | 13 | 21 | 19
Not completed — Lack of Efficacy | 5 | 4 | 8 | 10 | 20
Not completed — Adverse Event | 21 | 22 | 16 | 14 | 21
Not completed — Site termination/COPD exacerbation/other | 10 | 8 | 9 | 9 | 14

BASELINE CHARACTERISTICS:
Population: Safety population comprising all patients randomized to a treatment group who received at least 1 dose of double-blind investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo | Total
Number analyzed (Participants) | 335 | 333 | 337 | 332 | 332 | 1669
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.9) | 63.9 (9.2) | 64.4 (8.7) | 63.7 (8.7) | 63.5 (8.9) | 63.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 146 | 149 | 163 | 157 | 782
  Male | 168 | 187 | 188 | 169 | 175 | 887

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 1-hour Morning Post-dose Forced Expiratory Volume in One Second (FEV1)
Time Frame: Week 24 of treatment
Population: ITT Population defined as all randomized patients who took at least one administration of study medication and had a baseline and at least one post-baseline FEV1 assessment
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 335 | 333 | 337 | 332 | 331
Liters | 0.247 (0.013) | 0.226 (0.013) | 0.139 (0.013) | 0.165 (0.013) | -0.037 (0.014)
Statistical Analysis 1: Comparison: Aclidinium/Formoterol 400/12 μg vs Aclidinium 400 μg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment, sex, smoking-status, visit and group-by-visit as factors; screening pre- and post-bronchodilator FEV1, age and baseline FEV1 as covariates; Least squares mean difference = 0.108, 95% CI 2-sided [0.073 to 0.144], Standard Error of Mean 0.018
Statistical Analysis 2: Comparison: Aclidinium/Formoterol 400/6 μg vs Aclidinium 400 μg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.087, 95% CI 2-sided [0.052 to 0.123], Standard Error of Mean 0.018

2. Primary Outcome: Change From Baseline in Morning Trough Forced Expiratory Volume in One Second (FEV1)
Time Frame: Week 24 of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 335 | 333 | 337 | 332 | 331
Liters | 0.095 (0.012) | 0.076 (0.012) | 0.066 (0.012) | 0.050 (0.012) | -0.035 (0.013)
Statistical Analysis 1: Comparison: Aclidinium/Formoterol 400/12 μg vs Formoterol 12 μg; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.045, 95% CI 2-sided [0.011 to 0.079], Standard Error of Mean 0.017
Statistical Analysis 2: Comparison: Aclidinium/Formoterol 400/6 μg vs Formoterol 12 μg; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.026, 95% CI 2-sided [-0.008 to 0.060], Standard Error of Mean 0.017

3. Secondary Outcome: Change in Transition Dyspnea Index (TDI) Focal Score
Description: The TDI measures the change from baseline in severity of breathlessness in symptomatic patients. The TDI contains a rating for 3 categories (functional impairment, magnitude of task, magnitude of effort).TDI scale ranges from -3 (major deterioration) to +3 (major improvement) including a 0 score to indicate "no change". The 3 categories are added to obtain a focal score ranging from -9 (including 0) to +9.
Time Frame: Week 24 of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 335 | 333 | 337 | 332 | 331
Scores on a scale | 2.017 (0.203) | 1.977 (0.199) | 1.558 (0.201) | 1.522 (0.201) | 0.582 (0.216)
Statistical Analysis 1: Comparison: Aclidinium/Formoterol 400/12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment group, sex, smoking-status, visit, and treatment group-by-visit as factors; visit, age baseline BDI/SGRQ as covariates; Least squares mean difference = 1.436, 95% CI 2-sided [0.854 to 2.018], Standard Error of Mean 0.297
Statistical Analysis 2: Comparison: Aclidinium/Formoterol 400/6 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Least squares mean difference = 1.395, 95% CI 2-sided [0.818 to 1.972], Standard Error of Mean 0.294

4. Secondary Outcome: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Total Score
Description: St George's Respiratory Questionnaire (SGRQ) measures COPD-specific health outcomes and consists of 2 parts with 3 dimension scores (a symptom score and an activity and impacts score). SGRQ total score is the sum of these scores and ranges from 0 (best health status) to 100 (worst health status).
Time Frame: Week 24 of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Number analyzed (Participants) | 335 | 333 | 337 | 332 | 331
Scores on a scale | -6.568 (0.740) | -5.942 (0.728) | -6.438 (0.738) | -4.701 (0.742) | -2.215 (0.779)
Statistical Analysis 1: Comparison: Aclidinium/Formoterol 400/12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Least squares mean difference = -4.353, 95% CI 2-sided [-6.462 to -2.244], Standard Error of Mean 1.075
Statistical Analysis 2: Comparison: Aclidinium/Formoterol 400/6 μg vs Placebo; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Least squares mean difference = -3.728, 95% CI 2-sided [-5.819 to -1.637], Standard Error of Mean 1.066

ADVERSE EVENTS:
Time Frame: Week 26 ± 5 days
Description: Safety population comprised all patients randomized to a treatment group who received at least 1 dose of double-blind investigational treatment.
Arm/Group | Aclidinium/Formoterol 400/12 μg | Aclidinium/Formoterol 400/6 μg | Aclidinium 400 μg | Formoterol 12 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 19/335 | 18/333 | 17/337 | 15/332 | 12/332
Other Adverse Events (participants affected / at risk) | 63/335 | 65/333 | 57/337 | 74/332 | 58/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium/Formoterol 400/12 μg (N=335) | Aclidinium/Formoterol 400/6 μg (N=333) | Aclidinium 400 μg (N=337) | Formoterol 12 μg (N=332) | Placebo (N=332)
Pneumonia (Infections and infestations) | 2 | 1 | 1 | 3 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 1 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 1 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium/Formoterol 400/12 μg (N=335) | Aclidinium/Formoterol 400/6 μg (N=333) | Aclidinium 400 μg (N=337) | Formoterol 12 μg (N=332) | Placebo (N=332)
Nasopharyngitis (Infections and infestations) | 16 | 17 | 12 | 22 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 7 | 10 | 12
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 51 | 49 | 57 | 53 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Investigator will be subject to mutual agreement between the investigator and sponsor.